CLINICAL TRIAL: NCT00719836
Title: A Phase 1/2 Study of SB1518 for the Treatment of Advanced Myeloid Malignancies
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: S*BIO (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SB1518-2007-001
Record Dates: First submitted 2008-07-20; First posted 2008-07-22 (Estimated); Last update posted 2012-04-20 (Estimated); Status verified 2012-04

CONDITIONS: Acute Myelogenous Leukemia; Chronic Myelogenous Leukemia; Chronic Myelomonocytic Leukemia; Myelodysplastic Syndromes; Myelofibrosis
Keywords: SB1518; Chronic Idiopathic Myelofibrosis; JAK2 Inhibitor
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Leukemia, Myelomonocytic, Chronic; Myelodysplastic Syndromes; Primary Myelofibrosis | interventions — 11-(2-pyrrolidin-1-ylethoxy)-14,19-dioxa-5,7,26-triazatetracyclo(19.3.1.1(2,6).1(8,12))heptacosa-1(25),2(26),3,5,8,10,12(27),16,21,23-decaene

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: SB1518 — SB1518 taken orally daily for 28 consecutive days in a 28-day cycle

SUMMARY:
This study consists of two phases: the first portion of the study is a Phase 1 dose escalation study to determine the maximum tolerated dose and the dose limiting toxicities of SB1518 when given as a single agent orally once daily in subjects with advanced myeloid malignancies; the second portion of the study is a Phase 2 study to define the efficacy and safety profile of single-agent SB1518 at the recommended dose in subjects with chronic idiopathic myelofibrosis (CIMF).

ELIGIBILITY:
Inclusion Criteria

* During the dose escalation phase: subjects with histologically confirmed myeloid malignancy who have failed standard therapies or are not candidates for palliative therapies. This includes the following:

  * Subjects with Acute Myelogenous Leukemia (AML)
  * Subjects with Chronic Myelogenous Leukemia (CML) in accelerated phase
  * Subjects with Chronic Myelogenous Leukemia (CML) in blast crisis
  * Subjects with high-risk Myelodysplastic Syndromes (MDS) or Chronic Myelomonocytic Leukemia (CMML)
  * Subjects with Advanced Myelofibrosis (MF)
  * In Phase 2, subjects with CIMF (as well as post ET/PV MF)
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* All men of reproductive potential and women of child-bearing potential must agree to practice effective contraception during the entire study period and for one month after the last study treatment, unless documentation of infertility exists. Additionally, women of child-bearing potential must have a negative pregnancy test within 14 days prior to the first dose of study drug
* Able to understand and willing to sign the informed consent form

Exclusion Criteria

* Subjects with Chronic Myelogenous Leukemia (CML) in chronic phase;
* Uncontrolled inter-current illness including, but not limited to, ongoing active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements as judged by treating physician. Subjects receiving antibiotics for infections that are under control may be included in the study;
* Concurrent malignancy, except those subjects with early stage squamous cell carcinoma of the skin, basal cell carcinoma of the skin, or cervical intraepithelial neoplasia are eligible for the study;
* Known HIV-positive (such subjects are at increased risk of lethal infections when treated with potentially marrow-suppressive therapy);
* Known active hepatitis A, B, or C;
* Women who are pregnant or lactating.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2008-08; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Phase 1: To establish the maximum tolerated dose of SB1518 as a single agent when administered orally daily in subjects with advanced myeloid malignancies | Throughout the study
Phase 2: to assess the clinical benefit rate in subjects with CIMF who are treated with SB1518 at the recommended dose. | Throughout the study

SECONDARY OUTCOMES:
Assess the safety and tolerability of SB1518, administered once daily in subjects with advanced myeloid malignancies | Throughout the study
Assess the pharmacokinetic and pharmacodynamic profile of SB1518 | Throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: Srdan Verstovsek, M.D, Ph.D, Principal Investigator — M.D. Anderson Cancer Center; H. Joachim Deeg, M.D, Principal Investigator — Fred Hutchinson Cancer Center; Olatoyosi M. Odenike, M.D., Principal Investigator — The University of Chicago Hospitals
Locations (3):
- United States (3):
  - The University of Chicago Hospitals, Chicago, Illinois
  - MD Anderson Cancer Center, Houston, Texas
  - Fred Hutchinson Cancer Center, Seattle, Washington

REFERENCES:
- [Derived] Verstovsek S, Odenike O, Singer JW, Granston T, Al-Fayoumi S, Deeg HJ. Phase 1/2 study of pacritinib, a next generation JAK2/FLT3 inhibitor, in myelofibrosis or other myeloid malignancies. J Hematol Oncol. 2016 Dec 8;9(1):137. doi: 10.1186/s13045-016-0367-x. PMID 27931243